CLINICAL TRIAL: NCT05082506
Title: Effect of Acupressure on Pain, Anxiety and Vital Signs in Patients With Coronary Angiography: A Randomized Controlled Study
Brief Title: Effect of Acupressure on Pain, Anxiety and Vital Signs in Patients With Coronary Angiography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Selda Bal, SENİOR İNSTRUCTİON, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 41/21
Record Dates: First submitted 2021-09-08; First posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Pain; Anxiety; Vital Signs; Coronary Angiography
Keywords: pain; anxiety; vital signs; coronary angiography
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: Since the patients who will be included in the study are not known in advance, the patients will be randomized by the statistician using GraphPad software 3 and the block randomization technique, in order to assign the same number of participants to each group before the study, and will be divided into groups A, B, and C.
Who Masked: Participant
Masking Description: As a result of the draw, group A was determined as acupressure, group B as sham acupressure and group C as the control group. Since pressure will be applied to the pressure points of the patients in the acupressure and sham group included in the study, the sham (placebo) acupressure and acupressure groups will be blinded, since the patients do not know whether acupressure or sham acupressure is applied. The control group and the researcher cannot be blinded due to the nature of the research.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupressure Group (Experimental): Applicable to the acupressure group; Heart meridian 7th point (HT7), large intestine meridian 4th point (LI4) and pericardium 6th point (PC6), a total of three points will be applied. Afterwards, sequential (breathing rhythm) compressions will be applied to the determined acupressure points by the researcher without lifting the finger, taking into account the pain threshold of the individual who is applied with the thumb, with 10 seconds of pressure for two seconds of relief. Since the symmetry of the selected three different points on the other extremity will also be applied, a total of 12 minutes of compression will be applied to each point, provided that it is two minutes. Depending on the preparation and compression time on each point, the session duration of each patient will be approximately 16 minutes.
  Interventions: Behavioral: Acupressure
- Sham Group (Placebo Comparator): n the acupressure application to the Sham group, pressure will be exerted on the bone region where the meridians do not pass, parallel to the HT7, LI4, PC6 and points (approximately 1-1.5 cm away) (Figure 4). Before the application, the acupressure points will be heated for about 20 seconds and the tissue sensitivity will be reduced by rubbing and they will be made ready for the acupressure application. Afterwards, the acupressure points determined will be pressed with the thumb by the researcher with a lower intensity than the normal application pressure for two minutes. Similar to the acupressure group, the sham group will be applied to symmetrical points. In this direction, a session will last 16 minutes for each patient, as in the acupressure group, together with the duration of the pre-procedure preparation and applications.
  Interventions: Behavioral: Acupressure
- Control Group (No Intervention): Patients in the control group will not receive any intervention.

INTERVENTIONS:
Behavioral: Acupressure — Afterwards, sequential (breathing rhythm) compressions will be applied to the determined acupressure points by the researcher without lifting the finger, taking into account the pain threshold of the individual who is applied with the thumb, with 10 seconds of pressure for two seconds of relief.
  Arms: Acupressure Group; Sham Group

SUMMARY:
The study was planned to determine the effect of acupressure on pain, anxiety and vital signs of patients with coronary angiography. Acupressure application was carried out by the responsible researcher, who is certified on this subject, by TRNC Dr. In the Cardiology Service of Burhan Nalbantoğlu Hospital, patients who have undergone angiography will be applied and measurements will be made before mobilization after their informed consent is obtained.

DETAILED DESCRIPTION:
In this study, it is aimed to raise awareness for the use of painless, painless, economical, side-effect-free and easy-to-apply acupressure in nursing care in order to increase patient comfort by relieving pain and anxiety of patients during mandatory bed rest after coronary angiography. In addition, our study is important in terms of providing new information with a high level of evidence and providing a source for other studies on this subject.

Objective: The study was planned to determine the effect of acupressure on pain, anxiety and vital signs of patients with coronary angiography.

Hypothesis 1 H0: There is no difference in Visual Analog Scale mean scores between the acupressure group, the sham (pseudo-acupressure) group, and the control group.

H1: There is a difference in Visual Analog Scale mean scores between the acupressure group, the sham (pseudo-acupressure) group, and the control group.

Hypothesis 2 H0: There is no difference between the Spielberger State Anxiety Inventory mean scores between the acupressure group, the sham (pseudo-acupressure) group, and the control group.

H1: There is a difference between the Spielberger State Anxiety Inventory mean scores between the acupressure group, the sham (pseudo-acupressure) group, and the control group.

Hypothesis 3 H0: There is no difference in Systolic Blood Pressure between the acupressure group, the sham (false acupressure) group and the control group.

H1: There is a difference in Systolic Blood Pressure between the acupressure group, the sham (false acupressure) group and the control group.

Hypothesis 4 H0: There is no difference in Diastolic Blood Pressure between the acupressure group, the sham (false acupressure) group and the control group.

H1: There is a difference in Diastolic Blood Pressure between the acupressure group, the sham (false acupressure) group and the control group.

Hypothesis 5 H0: There is no difference in Heart Rate between the acupressure group, the sham (false acupressure) group and the control group.

H1: There is a difference between the acupressure group, the sham (false acupressure) group and the control group in terms of Heart Rate.

Hypothesis 6 H0: There is no difference in Respiration Rate between the acupressure group, the sham (false acupressure) group and the control group.

H1: There is a difference between the acupressure group, the sham (false acupressure) group and the control group in terms of Respiration Rate.

Hypothesis 7 H0: There is no difference in Cortisol Level between the acupressure group, the sham (false acupressure) group and the control group.

H1: There is a difference between the acupressure group, the sham (false acupressure) group and the control group in terms of Cortisol Level.

"Personal Information Form, "Spielberger State Anxiety Scale", "Visual Analogue Scale" and "Vital Signs Follow-up Form" will be administered to all patients (acupressure, sham acupressure and control groups) included in the study (1. "Spielberger State Anxiety Inventory", "After the measurement, half an hour after applying acupressure to the points determined for both groups (2nd measurement), two hours later (3rd measurement) and just before mobilization (4th measurement)," "Visual Analogue Scale" and "Vital Signs Follow-up Form" will be applied again.

It was created by the researcher to track the cortisol level. It is designed to include a total of 2 measurements (pre/post acupressure).

ELIGIBILITY:
Inclusion Criteria:

* First time coronary angiography performed
* Coronary angiography performed from the femoral region,
* over the age of 18,
* Willing to participate in the research,
* Able to understand and speak Turkish,
* Open to communication,
* Planned (non-urgent) coronary angiography
* No complications after angiography
* Stent etc. during angiography. no other attempt has been made
* No deformity or lesion in the areas where acupressure will be applied
* Not taking sedatives or pain relievers 5 hours before the angiography procedure,
* No acupressure experience
* Not diagnosed with anxiety disorder and not receiving medical treatment
* Not diagnosed with depression and not receiving medical treatment
* No chronic pain
* Patients without mental illness.

Exclusion Criteria:

* - Previous coronary angiography
* Coronary angiography from the femoral region is not performed,
* under the age of 18,
* pregnant,
* Those who do not agree to participate in the research,
* Can't understand or speak Turkish,
* Unable to communicate
* Unplanned (urgent) Coronary angiography Patients
* Any complications after angiography
* Stent etc. during angiography. another attempt has been made
* Any deformity or lesion in the areas where acupressure will be applied,
* Those who took sedatives or painkillers 5 hours before the angiography procedure,
* Experience with acupressure
* Anxiety disorder and receiving treatment,
* Diagnosed with depression and receiving treatment,
* Having chronic pain,
* Patients with mental disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 105 (Estimated)
Dates: Start 2021-12-15 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Spielberger State Anxiety Scale | 6 month
  The scale consists of 20 statements. The total score can range from 20 to 80. A high score indicates a high level of anxiety, and a low score indicates a low level of anxiety.

SECONDARY OUTCOMES:
Visual Pain Scale | 6 month
  It is a scale that is evaluated by individuals by making markings on a horizontal or vertical line of 10 cm or 100 mm, one end of which indicates that the patient is very good and the other end is very bad.

CONTACTS AND LOCATIONS:
Locations (1):
- Selda Bal, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP, ICF, CSR

REFERENCES:
- [Result] Virani SS, Alonso A, Aparicio HJ, Benjamin EJ, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Cheng S, Delling FN, Elkind MSV, Evenson KR, Ferguson JF, Gupta DK, Khan SS, Kissela BM, Knutson KL, Lee CD, Lewis TT, Liu J, Loop MS, Lutsey PL, Ma J, Mackey J, Martin SS, Matchar DB, Mussolino ME, Navaneethan SD, Perak AM, Roth GA, Samad Z, Satou GM, Schroeder EB, Shah SH, Shay CM, Stokes A, VanWagner LB, Wang NY, Tsao CW; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2021 Update: A Report From the American Heart Association. Circulation. 2021 Feb 23;143(8):e254-e743. doi: 10.1161/CIR.0000000000000950. Epub 2021 Jan 27. PMID 33501848
- [Result] Sharif F, Najafi Kalyani M, Ahmadi F, Iman MT. In the shadow of perceived threat: The live experience of Iranian patients candidate for undergoing coronary angiography. J Vasc Nurs. 2018 Sep;36(3):140-144. doi: 10.1016/j.jvn.2018.04.004. Epub 2018 Jun 7. PMID 30139451
- [Result] Caldwell PH, Arthur HM, Natarajan M, Anand SS. Fears and beliefs of patients regarding cardiac catheterization. Soc Sci Med. 2007 Sep;65(5):1038-48. doi: 10.1016/j.socscimed.2007.04.010. Epub 2007 May 15. PMID 17507132
- [Result] Shoulders-Odom B. Management of patients after percutaneous coronary interventions. Crit Care Nurse. 2008 Oct;28(5):26-41; quiz 42. No abstract available. PMID 18827085
- [Result] Fereidouni Z, Kameli Morandini M, Najafi Kalyani M. The efficacy of interventions for back pain in patients after transfemoral coronary angiography: A rapid systematic review. J Vasc Nurs. 2019 Mar;37(1):52-57. doi: 10.1016/j.jvn.2018.11.002. Epub 2018 Dec 17. PMID 30954199
- [Result] Tolentino JC, Schmidt JJ, Schmidt GJ, Mesquita CT, Schmidt SL. Mental Stress-Induced Myocardial Ischemia Related to Generalized Anxiety Disorder in a Patient With Acute Coronary Syndrome and Normal Coronary Arteries. Clin Nucl Med. 2016 Nov;41(11):e487-e490. doi: 10.1097/RLU.0000000000001348. PMID 27607164
- [Result] Au DW, Tsang HW, Ling PP, Leung CH, Ip PK, Cheung WM. Effects of acupressure on anxiety: a systematic review and meta-analysis. Acupunct Med. 2015 Oct;33(5):353-9. doi: 10.1136/acupmed-2014-010720. Epub 2015 May 22. PMID 26002571
- [Result] Khoram B, Yoosefinejad AK, Rivaz M, Najafi SS. Investigating the Effect of Acupressure on the Patients' Anxiety Before Open-Heart Surgery: A Randomized Clinical Trial. J Acupunct Meridian Stud. 2020 Dec;13(6):169-173. doi: 10.1016/j.jams.2020.11.001. Epub 2020 Nov 24. PMID 33242637
- [Result] Sharifi Rizi M, Shamsalinia A, Ghaffari F, Keyhanian S, Naderi Nabi B. The effect of acupressure on pain, anxiety, and the physiological indexes of patients with cancer undergoing bone marrow biopsy. Complement Ther Clin Pract. 2017 Nov;29:136-141. doi: 10.1016/j.ctcp.2017.09.002. Epub 2017 Sep 5. PMID 29122251